CLINICAL TRIAL: NCT01102842
Title: Unattended In-home Sleep Recording: A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 09-192-A
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Laboratory studies have found that insufficient sleep duration and impaired sleep quality are associated with disease risk, including obesity, diabetes and heart disease. The limitation to the laboratory studies is that they are conducted in artificial environments that do not reflect real-world behavior. Although the epidemiologic studies do reflect habitual behavior, the vast majority of them rely on self-reported measures of sleep, which are only moderately correlated with objective measures of sleep.. The next logical step in the examination of sleep's role in cardiometabolic health is to conduct objective, detailed measures of sleep in people's homes. This project is a pilot study that will develop ideal methodologies for recording sleep in the home environment. Because there is currently is a gap between laboratory models of sleep loss and real world conditions, the ultimate goal of this research is to expand our work on sleep and cardiometabolic health outside of the laboratory. Given the strong evidence for a link between impaired and insufficient sleep and increased disease risk, it is critical that we understand how people sleep in their daily lives and what factors can impact sleep. This project will record sleep in people's homes using ambulatory polysomnography recordings and wrist actigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Must have had a polysomnography recording at the University of Chicago.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers (18 years of age and older) who have had a polysomnography recording in the laboratory at the University of Chicago.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sleep Architecture | once
  Sleep architecture (stages) from polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Knutson, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States